CLINICAL TRIAL: NCT02707289
Title: Retrospective Collection of PillCam SB Movies for Capsule Transit Time Analysis (OCEAN Study)
Brief Title: Retrospective Collection of PillCam SB Movies
Acronym: OCEAN
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVGIBD0547
Record Dates: First submitted 2016-03-02; First posted 2016-03-14 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Inflammatory Bowel Disease, Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Up to two hundred un-identified PillCam SB movies will be collected from 2 clinical sites, during up to 3 years and transferred to Given Imaging. Demographical data and medical history will be collected. Capsule transit time in the different sections of the GI will be evaluated.

DETAILED DESCRIPTION:
Up to two hundred un-identified PillCam SB movies that were created between the year 2008 and the date the study was approved by the IRB, will be collected from 2 clinical sites, Sourasky and Sheba medical centers during up to 3 years and transferred to Given Imaging. Demographical data and medical history will be collected. Capsule transit time in the different sections of the GI will be evaluated by internal readers.

ELIGIBILITY:
Inclusion Criteria:

Videos collected from any PillCam SB procedure

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to two hundred un-identified PillCam SB movies that were created between the year 2008 and the date the study was approved by the IRB, will be collected
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Transit time in the different sections of the GI according to PillCam SB movies (minutes) | Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Eliakim, Prof., Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No